CLINICAL TRIAL: NCT03769753
Title: Trial Of IRE in Cholangiocarcinoma (TOnIC): Phase II
Brief Title: Trial of IRE in Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-489
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Results first posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Cholangiocarcinoma
Keywords: intraoperative use of IRE; 18-489
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center phase I study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- intraoperative use of IRE (Experimental): Patients with intraoperatively determined advanced unresectable PHC will be treated with IRE during the same surgical exploration session (N=20). Electrodes will be placed using ultrasound guidance. All electrodes will be placed by hepatopancreatobiliary surgeons with experience using IRE.
  Interventions: Device: IRE Device

INTERVENTIONS:
Device: IRE Device — For use in ablating soft tissue
  Other Names: The NanoKnife IRE device

SUMMARY:
The purpose of this study is to test any good and bad side effects of surgery using IRE to treat cancer of the bile duct.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Capable of providing written and oral informed consent in English
* Locally advanced disease based on preoperative work-up demonstrating that the tumor is unresectable due to portal vein, hepatic artery, and/or bile duct involvement, insufficient hypertrophy response of the future liver remnant after portal vein embolization, or patients not able to tolerate major liver surgery
* Found to be unresectable intraoperatively based on vascular, biliary, or lymph node (N2) involvement upon exploratory laparotomy
* Patients will be assessed for chemotherapy prior to treatment with IRE, but given the common problem of recurrent cholangitis, some patients will not be candidates for chemotherapy until after IRE is performed.

Exclusion Criteria:

* Locally advanced PHC eligible and accepted for liver transplantation evaluation
* PHC with > 5 cm extension along the common hepatic duct or common bile duct on preoperative imaging or intraoperative ultrasound
* Metastases to peritoneum, liver or other organs confirmed by percutaneous biopsy, staging laparoscopy or intraoperative frozen section
* Lymph node metastases beyond N2 stations, confirmed by intraoperative frozen sections or radiographic diagnosis
* History of cardiac disease:

  * Congestive heart failure (NYHA class >2)
  * Active Coronary Artery Disease (defined as myocardial infarction within 6 months prior to screening)
  * Cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker (beta blockers are permitted)
* Any implanted stimulation device (defined as implantable cardiac device and a pacemaker)
* Uncontrolled hypertension (blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen)
* Uncontrolled infections (> grade 2 NCI-CTC, version 3.0)
* Epilepsy
* Both narrowing (sclerosis) of the main portal vein and a reduced diameter of either the common hepatic artery, celiac trunk or superior mesenteric artery of >50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T. Peter Kingham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Basking Ridge (Consent and Follow up), Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth (Consent and Follow up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow up), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow up), Commack, New York
  - Memoral Sloan Kettering Westchester (Consent and Follow Up), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-up), Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative Use of IRE
Started | 8
Completed | 1
Not Completed | 7
Not completed — Not Treated | 6
Not completed — Inevaluable - No Evidence of Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Use of IRE
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 72 [64 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing a Clinically Relevant Complications
Description: defined as CTCAE (version 5.0) grade 3 or higher complications
Time Frame: within 30 days post-IRE
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Use of IRE
Number analyzed (Participants) | 8
Participants
  Number of participants with grade 3 or higher complications | 1
  Number of participants not evaluated for complications | 7

ADVERSE EVENTS:
Time Frame: within 30 days post-IRE
Arm/Group | Intraoperative Use of IRE
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Use of IRE (N=8)
Alkaline phosphatase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03769753/Prot_SAP_000.pdf